CLINICAL TRIAL: NCT00897247
Title: Early Detection Biomarkers for Mesothelioma Among Asbestos and Vermiculite Exposed Populations
Brief Title: Biomarkers to Detect Mesothelioma Early in Patients Exposed to Asbestos or Vermiculite
Status: Completed | Type: Observational
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000518348; P30CA022453 (NIH); WSU-2006-057; WSU-HIC-094806MP2F
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Malignant Mesothelioma; Pulmonary Complications
Keywords: malignant mesothelioma; pulmonary complications
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Microarray Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis
Genetic: protein expression analysis
Genetic: proteomic profiling
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of body fluid and blood from patients who have been exposed to asbestos or vermiculite in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking for biomarkers to detect mesothelioma early in patients exposed to asbestos or vermiculite.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify patients with known asbestos exposure at early stages of disease development (i.e., indolent premalignant pleural plaques and fibrosis vs malignant pleural mesothelioma).
* Determine the expression levels of tumor-associated proteins in these patients.
* Analyze samples of serum and pleural effusions obtained from these patients.
* Determine the proteomic profile of samples obtained from these patients.
* Determine the molecular mechanisms associated with the regulation of the extracellular matrix microenvironment proteins (e.g., osteonectin, intelectin, or matrix metalloproteins) involved in disease onset and progression.

OUTLINE: This is a multicenter study.

Patients undergo collection of body cavity fluid, including pleural effusion, and blood. Specimens, including fresh frozen malignant pleural mesothelioma tumor tissue, if available, are analyzed for proteomic profile, gene expression profile, and tumor-associated protein expression levels.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Exposure to vermiculite or asbestos insulation

  * Symptomatic or nonsymptomatic exposure-related disease
* Seen at a clinic in Libby, Montana (CARD Clinic) or Michigan (COEM)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2007-01; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Identification of potential drug targets for therapeutic strategies to treat asbestos fiber-related diseases | At time of analysis

CONTACTS AND LOCATIONS:
Overall Officials: Anil Wali, PhD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States